CLINICAL TRIAL: NCT03668080
Title: Burnout Syndrome Among Medical Residents
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, matteo serenari, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: 105543
Record Dates: First submitted 2018-09-09; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Burnout Syndrome
Keywords: burnout; residents; surgical residents
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- surgical residents: Surgical specialties included general surgery, plastic surgery, urology, vascular surgery, obstetrics and gynecology, orthopedic surgery, pediatric surgery, cardiothoracic surgery and otolaryngology.
- non-surgical residents: Non-surgical specialties included cardiology, rheumatology, neurology, pulmonary disease, endocrinology, nuclear medicine, pediatrics, psychiatry, internal medicine, oncology, nephrology, hygiene and preventive medicine, anesthesiology, child and adolescent psychiatry, radiology, radiation oncology, infectious disease, dermatology, pathology, microbiology, hematology, gastroenterology, geriatric medicine, medical genetics, sports medicine, occupational and environmental medicine.

SUMMARY:
Whether and to what extent burnout risk is actually higher in surgical specialties than in non-surgical specialties is still unknown. Little is also known about what factors are associated with burnout between surgical residents and non-surgical residents. In this context, the present study has a three-fold aim: 1) to measure the prevalence of burnout among a sample of Italian medical residents; 2) to contrast the prevalence of burnout and psychological distress in surgical residents and non-surgical residents, and 3) to identify the work-related factors associated with burnout between surgical residents and non-surgical residents.

DETAILED DESCRIPTION:
Surgical training is considered to be very stressful among residents and graduating medical students choose less often surgery for their career. To elaborate burnout prevention programs, the assessment of the prevalence of burnout during the early career stage of the surgeons and associated risk factors, becomes central.

Residents from the University of Bologna were asked to participate in an anonymous online survey. The residents completed a set of questions regarding their training schedule and three standardized questionnaires: 1) the Maslach Burnout Inventory, assessing the three dimensions of burnout: emotional exhaustion (EE), depersonalization (DP), and personal accomplishment (PA); 2) the Zung Self-Rating Depression scale; 3) the Psychosomatic Problems scale. High scores in either the EE or DP subscale categories predicted professional burnout.

ELIGIBILITY:
Inclusion Criteria:

* residents attending the University of Bologna

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the residents attending the University of Bologna in the academic year 2017/2018
Sampling Method: Non-Probability Sample
Enrollment: 679 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2017-11-05 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Maslach Burnout Inventory | 3 months
  a validated 22-item questionnaire that evaluates burnout in its three dimensions: emotional exhaustion (EE) depersonalization (DP) and personal accomplishment (PA). Responses are made on a 7-point Likert scale ranging from 0 ("never") to 6 ("daily").

SECONDARY OUTCOMES:
Zung Self-Rating Depression Scale | 3 months
  The level of depressive symptoms was measured using the 20-item Zung Self-Rating Depression Scale. Items responses rank from 1 ("none or little of the time") to 4 ("most or all of the time"), and the total score range from 20 to 80 points. A score of 50 and above indicated the presence of at least mild-moderate depressive symptoms.
Psychosomatic Problems Scale | 3 months
  Psychosomatic symptoms were measured using the Psychosomatic Problems Scale, which consists of 8 items: difficulty concentrating, sleep problems, headache, stomachache, tensions, lack of appetite, feeling sad, and dizziness. Responses are rated on a 5-point Likert scale, ranging from 1 ("never") to 5 ("always"). Participants answering "often" or "always" on an item are coded as having a psychosomatic symptom.

CONTACTS AND LOCATIONS:
Overall Officials: antonio d pinna, MD, Study Director — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- University of Bologna, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maslach C, Schaufeli WB, Leiter MP. Job burnout. Annu Rev Psychol. 2001;52:397-422. doi: 10.1146/annurev.psych.52.1.397. PMID 11148311
- [Derived] Serenari M, Cucchetti A, Russo PM, Fallani G, Mattarozzi K, Pinna AD, Colonnello V, Poggioli G, Cescon M. Burnout and psychological distress between surgical and non-surgical residents. Updates Surg. 2019 Jun;71(2):323-330. doi: 10.1007/s13304-019-00653-0. Epub 2019 Apr 2. PMID 30941702